CLINICAL TRIAL: NCT03031028
Title: The Study of Outpatient Ketogenic Diet on Seizure Rate, Nutritional Status and Some Biochemical Factors in Children and Adolescent With Refractory Epilepsy.
Brief Title: Effect of Outpatient Classic Ketogenic Diet in Epileptic Children and Adolescent.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94-03-161-30342
Record Dates: First submitted 2016-12-31; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-09

CONDITIONS: Refractory Epilepsy
Keywords: refractory epilepsy,; ketogenic diet; classic ketogenic diet; seizure rate; efficacy; epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ketogenic diet (Other): Ketogenic diet
  Interventions: Other: ketogenic diet

INTERVENTIONS:
Other: ketogenic diet — Ketogenic Diet is a high fat, low carbohydrate diet.

SUMMARY:
This study will consider the effectiveness of the ketogenic diet (high-fat, low-carbohydrate, and moderate protein) in treating epilepsy. Investigators enroll a group of eligible epileptic children and adolescent who have been referred from epilepsy center to our clinic and prescribe them ketogenic diet.

DETAILED DESCRIPTION:
This research will be done to observe efficacy, safety, and tolerability of the classic ketogenic diet (CKD) on an outpatient basis without fasting, caloric and fluid restriction in children with and adolescents with intractable epilepsy.

30 children and adolescents with intractable epilepsy based on inclusion and exclusion criteria have been enrolled in the study, Investigators prescribe them classic ketogenic diet. Efficacy of the diet will be assessed through seizure rates, number of anti-epileptic drug used by the patients, and EEG changes. Seizure frequency will be assessed by seizure record diary that is filled out by family of the patients and will be compared with data that will be taken at 1, 3 months after start of the diet. EEG will be taken at baseline and 3 months after start of the diet. Patients will be reviewed at 1, 3 months after start of the diet at outpatient clinic. Intolerances and Complications will be documented at each clinic visits and via telephone calling during clinic visits intervals to evaluate tolerability and safety of the KD. For close monitoring of the complications along with blood tests and urinalysis Investigators will do echocardiography and renal ultrasound at baseline and 3 months after start of the diet. Laboratory values will be assessed at baseline and 3 months after start of the diet. Also, nutritional status and growth of children will be assessed at baseline and 1, 3 months after start of diet.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1-18 years,
* The patient has tried at least 3 different AED:s including one combination with two or more different AED:s.
* The parents are willing to include their child in the study after written and verbal information.
* Patients with all types of epilepsy can be included.
* The patient is submitted to our epilepsy center.

Exclusion Criteria:

* The patient has a medical condition, for example a metabolic disease, where ketogenic diet is contraindicated.
* The patient's nutritional status is not good enough or intake of fluid is to small to permit treatment with ketogenic diet.
* No history of hyperlipidemia
* No history of renal stones
* No previous treatment with ketogenic diet
* Beta-oxidation defects - medium-chain acyl dehydrogenase deficiency (MCAD), long-chain acyl dehydrogenase deficiency (LCAD), short-chain acyld dehydrogenase deficiency (SCAD), long-chain 3-hydroxyacyl-coenzyme A (CoA) deficiency, and medium-chain 3- hydroxyacyl-CoA deficiency.
* The family is expected to have compliance problems with treatment and/or seizure registration

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
seizure rate | 3 months
  The information will be obtained through seizure diary

SECONDARY OUTCOMES:
Height | Before and after 1 and 3 months on the classical KD.
  Height of the participants will be assessed by stadiometer and Unit for height is cm.
Investigating side effects | After 3 months on the classical KD
  Side effects will be obtained via parents' reports.
serum Triglyceride | Before and after 3 months on the classical KD
  serum Triglyceride will be assessed. Units for serum TG, is mg/dl.
Weight | Before and after 1 and 3 months on the classical KD.
  Weight of the participants will be assessed by seca scale and Unit for weight is kilogram.
serum Cholesterol, | Before and after 3 months on the classical KD
  serum Cholesterol will be assessed. Units for serum Cholesterol is mg/dL.
serum LDL-Cholesterol | Before and after 3 months on the classical KD.
  serum LDL-Cholesterol will be assessed. Units for serum LDL-C is mg/dL.
serum HDL-Cholesterol | Before and after 3 months on the classical KD
  serum HDL-Cholesterol will be assessed. Units for serum HDL-C is mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Mahmoudi, MD, PHD, Study Director — Tehran university of medical science, school of Nutritional science and Dietetics
Locations (1):
- Tehran university of medical science, school of nutritional science and dietetics, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided